CLINICAL TRIAL: NCT06262100
Title: Clinical Investigation to Evaluate the Lubricating Performance of Carragelose Containing Eye Drops in Patients Diagnosed with Mild-to-moderate Dry Eye Disease
Brief Title: Lubricating Effectiveness of Carragelose Eye Drops in Patients Affected by Mild to Moderate Dry Eye
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Marinomed Biotech AG (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EYL_23_01
Record Dates: First submitted 2024-01-31; First posted 2024-02-15 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-12

CONDITIONS: Dry Eye Syndromes
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Carragelose (Other): Treatment with Carragelose containing eye drops
  Interventions: Device: Carragelose

INTERVENTIONS:
Device: Carragelose — Application of Carragelose containing eye drops

SUMMARY:
Patients suffering from dry eye syndrom will treat their eyes with Carragelose® eye drops three times a day for 28 days. Before, in the middle and at the end of the treament period patients will be exposed to adverse conditions to challenge dry eye symptoms. Patient will record their occular symptoms and ophthalmic examinations will be performed by an ophthalmologist. Differences between before and after treatment will be assessed.

DETAILED DESCRIPTION:
The objective is to evaluate the safety and performance of Carragelose®-containing eye drops in treating symptoms and signs of dry eye syndrom.

Patients will treat their eyes with one eye drop three times a day for 28 days. Baseline assessment will be performed after normal controlled environment and after adverse controlled environment. At the end of investigation ocular symptoms and ocular sign will be assessed after normal controlled environment and after adverse controlled environment. Differences between baseline and end of investigation will be evaluated for efficacy analysis.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients (aged ≥ 18 years) from any sex or gender who provide written informed consent to participate.
2. Diagnosis of DED by an ophthalmologist having DED-related symptoms lasting at least 3 months.
3. Mild-to-moderate DED as defined above.
4. Patients who do not use or can do without the use of contact lenses from at least 7 (±2) days before the Inclusion visit (Visit 2) and throughout the entire study period.
5. Patients able to administer the study eye drops themselves in both eyes for the intended duration of the study (28 days).
6. Patients willing not to use any other eye drops during the entire study period.
7. Women with childbearing potential must commit to using effective methods of contraception during the entire study period and have a negative result on a pregnancy test at the Screening visit.

Exclusion Criteria:

1. Patients with known hypersensitivity, allergy, or intolerance to the IP or any of its components.
2. Patients with any ocular surface disease or condition other than DED.
3. Patients with any other active ocular inflammatory disease or condition, glaucoma or who have received any ocular surgery during the last 6 months.
4. Patients who have received lacrimal punctum occlusion during the previous month, or in whom it is planned during the study period.
5. Patients with any of the following seriousness criteria:

   * fluorescein corneal staining score ≥ 4 in the Oxford scale;
   * lissamine green conjunctival staining score ≥ 4 in the Oxford scale;
   * Schirmer test score < 2 mm;
   * fluorescein TBUT = 0 seconds.
6. Patients receiving any other topical ocular medication, such as non-steroidal anti-inflammatory drugs, etc. within 30 days of inclusion (Visit 2).
7. Patients with clinically relevant or uncontrolled systemic diseases (except for controlled Sjögren syndrome) during the last 3 months that may interfere with study assessments or results.
8. Patients requiring or who have received topical ocular treatment with calcineurin inhibitors (such as cyclosporin or tacrolimus) during the last 12 weeks, corticosteroids during the last 4 weeks, blood derivatives (such as autologous/allogeneic serum, platelet-rich plasma, plasma rich in growth factors or umbilical cord-derived plasma), insulin or amniotic membrane preparations during the last week, during the last month before the Inclusion visit (Visit 2).
9. Patients who have received treatment with any ocular lubricant after the Screening visit (Visit 1) other than the one specified in the protocol (Hydrabak).
10. Patients who have started systemic treatments that may affect DED signs or symptoms, ocular surface or vision, during the last 3 months or if a change in the dose of such treatments is expected during the study.
11. Inability to follow the study procedures, including attending all site visits, tests, and examinations.
12. Mental incapacity that precludes adequate understanding or cooperation.
13. Patients currently participating or who have participated in another investigational study during the last 30 days.
14. Pregnant or breastfeeding women.
15. Patients who, according to the investigator's criteria, are not suitable to participate in the study or comply with the study protocol.

    -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2024-01-15 (Actual); Primary Completion 2024-07-30 (Actual); Study Completion 2024-07-30 (Actual)

PRIMARY OUTCOMES:
Change in dry eye symptoms | 28 days
  Composite score on dry eye related ocular symptoms collected through numerical rating scales (NRS) for foreign body sensation, burning/stinging, itching, pain, sticky feeling, blurred vision, and photophobia.

SECONDARY OUTCOMES:
Responder analysis | 28 days
  Patient responder rates evaluated as per the Numeric rating scale (0 to 10) scores.

CONTACTS AND LOCATIONS:
Overall Officials: Margarita Calogne, PhD, Principal Investigator — IOBA, University of Valladolid
Locations (1):
- IOBA,Ocular Surface Research Group, University of Valladolid, Valladolid, Spain

IPD SHARING:
Plan to Share IPD: No